CLINICAL TRIAL: NCT00232128
Title: Protocol for Radiofrequency Ablation of Pulmonary Neoplasms
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Oncology Specialties, Alabama (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCI LUN 02
Record Dates: First submitted 2005-10-03; First posted 2005-10-04 (Estimated); Last update posted 2007-01-12 (Estimated); Status verified 2006-05

CONDITIONS: Pulmonary Neoplasms
MeSH Terms: conditions — Lung Neoplasms

INTERVENTIONS:
Procedure: Radiofrequency Ablation of pulmonary neoplasms

SUMMARY:
This research trial involves the development of a new treatment for lung tumors. It is for patients whose tumor cannot be surgically removed, have refused surgery, or the tumor has not responded well to other forms of treatment. This treatment uses a needle probe to deliver energy into the lung tumor. This probe is placed utilizing a CT scan image. The energy heats the tumor causing tumor cell death.

ELIGIBILITY:
Inclusion Criteria: The patients enrolled in this study should be judged to have sufficient survival to benefit from control of local disease and include at least one of the following:

1. unresectable primary or metastatic lung tumors
2. may benefit from multiple modalities of therapy
3. chemotherapeutic or radiation oncologic options have been exhausted

Exclusion Criteria:

1. co-existing morbidities that preclude the use of surgery

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2003-06

CONTACTS AND LOCATIONS:
Overall Officials: Marshall T. Schreeder, M.D., Principal Investigator — Comprehensive Cancer Institute
Locations (1):
- Comprehensive Cancer Institute, Huntsville, Alabama, United States

REFERENCES:
- See also: Related Info — http://www.ccihsv.com